CLINICAL TRIAL: NCT00413192
Title: Phase II Study of E7389 Administered as an IV Bolus Infusion Day 1 and Day 8 Every 3 Weeks in Pre-Treated Patients With Advanced and/or Metastatic Soft Tissue Sarcoma
Brief Title: E7389 Administered as an IV Bolus Infusion Day 1 and Day 8 Every 3 Weeks in Pre-Treated Patients With Advanced and/or Metastatic Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7389-E044-207; 2005-004272-20 (EudraCT Number)
Record Dates: First submitted 2006-12-15; First posted 2006-12-19 (Estimated); Results first posted 2017-03-22 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-01

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — eribulin

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: E7389

INTERVENTIONS:
Drug: E7389 — 1.4 mg/m^2 administered as an intravenous (I.V.) bolus infusion on Days 1 and 8 of every 21 days.

SUMMARY:
The purpose of this study is to evaluate the therapeutic activity and safety of E7389 in patients with advanced/metastatic soft tissue sarcoma who have failed standard chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven advanced and/or metastatic malignant soft tissue sarcoma of high or intermediate grade, and of one of the following histologies (World Health Organization (WHO) classification 2002):

   * Leiomyosarcoma
   * Adipocytic (liposarcoma dedifferentiated, myxoid/round cell, pleomorphic, mixed-type not otherwise specified)
   * Synovial sarcoma
   * Other types of sarcoma, including:
   * Fibroblastic (adult fibrosarcoma, myxofibrosarcoma, sclerosing epithelioid fibrosarcoma).
   * So-called fibrohistiocytic (pleomorphic Malignant Fibrous Histiocytoma (MFH), giant cell "MFH", inflammatory "MFH")
   * Malignant glomus tumors.
   * Skeletal muscles (rhabdomyosarcoma, alveolar or pleomorphic) excluding embryonal rhabdomyosarcoma.
   * Vascular (epithelioid haemangioendothelioma, angiosarcoma).
   * Uncertain differentiation (synovial, epithelioid, alveolar soft part, clear cell, desmoplastic small round cell, extra-renal rhabdoid, malignant mesenchymoma, perivascular epithelioid cell tumor (PEComa), intimal sarcoma) excluding chondrosarcoma, Ewing tumors / Primitive neuroectodermal tumor (PNET)
   * Malignant peripheral nerve sheath tumors.
   * Malignant solitary fibrous tumors.
   * Undifferentiated soft tissue sarcomas not otherwise specified.
   * Other types of sarcoma (not listed as not eligible), if approved by the Study Coordinator (written or e-mail approval needed prior to registration).
   * The following tumor types are not eligible:
   * Embryonal rhabdomyosarcoma
   * Chondrosarcoma
   * Osteosarcoma
   * Ewing tumors / PNET
   * Gastro-intestinal stromal tumors (GIST)
   * Dermatofibrosarcoma protuberans
   * Inflammatory myofibroblastic sarcoma
   * Neuroblastoma
   * Malignant mesothelioma
   * Mixed mesodermal tumors of the uterus
2. Formalin fixed paraffin embedded tumor blocks and representative H/E (hematoxylin/eosin) slides must be available for histological central review. Histological central review is not required before treatment start but is mandatory within 10 days of registration. Local histopathological diagnosis will be accepted for entry into the study.
3. Relapsed, refractory and/or metastatic disease incurable by surgery or radiotherapy.
4. Evidence of objective progression within the last 6 months (RECIST) documented by measurements of disease, i.e. appearance of new lesions, increase of 20% in the sum of the diameters of measurable lesions, or progression of non measurable lesions to be confirmed by an external review, without other specific treatment since objective documentation of progression.
5. Presence of measurable disease, as defined by RECIST.
6. Patients must have received no more than one combination or two single agent chemotherapy regimens for advanced disease; (neo)adjuvant therapy is not counted towards this requirement.
7. No major surgery, hormonal therapy (other than replacement), chemotherapy or radiotherapy, immunotherapy or other investigational agent within the last 28 days and/or not recovered from prior therapy within the last 28 days. Use of erythropoietin is considered supportive care and is permitted.
8. Absence of brain or subdural metastases, unless patient has completed local therapy and has discontinued the use of corticosteroids for this indication for at least 4 weeks before starting treatment with E7389. Any signs (e.g., radiologic) and/or symptoms of brain metastases must be stable for at least 4 weeks.
9. Absence of pre-existing neuropathy > Grade 2
10. At least 18 years of age.
11. WHO performance status 0 or 1.
12. Adequate bone marrow function (absolute neutrophil count >1.5 x 109/L, platelets >100 x 109/L)
13. Adequate hepatic function (bilirubin < 1.5 mg/mL or 25 µmol/L, SGOT/AST and SGPT/ALT <= 3 x UNL or < 5 x UNL in patients with liver metastases).
14. Adequate renal function: serum creatinine < 2.0 mg/dl or 177 µmol/l or calculated (Cockcroft and Gault formula) creatinine clearance > 40 ml/min.
15. Women should either not be of childbearing potential (having had a hysterectomy, a bilateral oophorectomy or bilateral tubal ligation, or be post-menopausal with a total cessation of menses of >1 year), or not be pregnant (negative serum pregnancy test at entry), should not be lactating, should agree to use contraceptive methods (with a documented failure rate < 1%, vasectomized partner sterile prior to trial entry and sole sexual partner or double-barrier contraception) while on treatment and during a period of 3 months after the end of treatment. Sexually active male participants must use barrier methods of contraception.
16. Before patient registration/randomization, written informed consent must be given according to International Conference on Harmonization/Good Clinical Practice (ICH/GCP), and national/local regulations.

Exclusion Criteria:

1. Prior history of malignancies other than sarcoma (except for basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or breast, or the patient has been free of any other malignancies for > 3 years).
2. Significant cardiovascular impairment (history of congestive heart failure > New York Heart Association (NYHA) grade II, unstable angina or myocardial infarction within the past six months, or serious cardiac arrhythmia).
3. Patients who are receiving anti-coagulant therapy with warfarin or related compounds, other than for line patency, and cannot be changed to heparin-based therapy, are not eligible. If a patient is to continue on mini-dose warfarin, then the prothrombin time (PT) / international normalized ratio (INR) must be closely monitored.
4. Severe/uncontrolled intercurrent illness/infection.
5. Patients with a known hypersensitivity to halichondrin B and/or halichondrin B chemical derivative.
6. Patients who participated in a prior E7389 clinical trial.
7. Patients without freedom (by the law or administrative decision), hospitalized without their consent (mental disability, upon legal request), admitted in medical or social establishment for other reasons than clinical research, with any psychological, familial, sociological, geographical condition potentially hampering compliance with the study protocol and follow-up schedule ; those conditions should be assessed with the patient before registration in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2007-01; Primary Completion 2012-06 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- Belgium (2):
  - Brussels
  - Leuven
- Denmark (2):
  - Aarhus
  - Herlev
- France (4):
  - Bordeaux
  - Lyon
  - Marseille
  - Villejuif
- Germany (6):
  - Bad Saarow
  - Dresden
  - Essen
  - Hanover
  - Mannheim
  - Tübingen
- Warsaw, Poland

REFERENCES:
- [Derived] Wiemer EAC, Wozniak A, Burger H, Smid M, Floris G, Nzokirantevye A, Sciot R, Sleijfer S, Schoffski P. Identification of microRNA biomarkers for response of advanced soft tissue sarcomas to eribulin: Translational results of the EORTC 62052 trial. Eur J Cancer. 2017 Apr;75:33-40. doi: 10.1016/j.ejca.2016.12.018. Epub 2017 Feb 16. PMID 28214655
- [Derived] Schoffski P, Ray-Coquard IL, Cioffi A, Bui NB, Bauer S, Hartmann JT, Krarup-Hansen A, Grunwald V, Sciot R, Dumez H, Blay JY, Le Cesne A, Wanders J, Hayward C, Marreaud S, Ouali M, Hohenberger P; European Organisation for Research and Treatment of Cancer (EORTC) Soft Tissue and Bone Sarcoma Group (STBSG). Activity of eribulin mesylate in patients with soft-tissue sarcoma: a phase 2 study in four independent histological subtypes. Lancet Oncol. 2011 Oct;12(11):1045-52. doi: 10.1016/S1470-2045(11)70230-3. Epub 2011 Sep 19. PMID 21937277

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 128 participants were enrolled. Of these 128 participants115 were eligible to continue in the study following reassessment of study eligibility in which 12 participants previously found eligible and began treatment, were then assessed as ineligible. One participant was not treated.
Groups:
- Adipocyte Tumors (ADI): Participants were administered 1.4 mg/m^2 eribulin mesilate by intravenous (IV) bolus infusion over 2 to 5 minutes on Days 1 and 8 every 21 days (21 Days = 1 Cycle) for as long as clinical benefit was sustained. The dose of study drug could have been reduced or discontinued during any treatment period, in accordance with toxicity modifications. Once the dose was reduced, it could not be increased at a later date.
- Leiomyosarcoma (LMS); Synovial Sarcoma (SYN); Other Types of Sarcoma (OTH): Participants were administered 1.4 mg/m^2 eribulin mesilate by intravenous (IV) bolus infusion over 2 to 5 minutes on Days 1 and 8 every 21 days (21 Days = 1 Cycle) for as long as clinical benefit was sustained. The dose of study drug could have been reduced or discontinued during any treatmeDnt period, in accordance with toxicity modifications. Once the dose was reduced, it could not be increased at a later date.
Period: Overall Study
Arm/Group | Adipocyte Tumors (ADI) | Leiomyosarcoma (LMS) | Synovial Sarcoma (SYN) | Other Types of Sarcoma (OTH)
Started | 37 | 40 | 19 | 32
Completed | 0 | 0 | 0 | 0
Not Completed | 37 | 40 | 19 | 32
Not completed — Disease progression | 26 | 31 | 16 | 25
Not completed — Toxicity | 3 | 2 | 2 | 2
Not completed — Withdrawal by Subject | 3 | 5 | 0 | 1
Not completed — Intercurrent illness | 0 | 0 | 0 | 1
Not completed — Intercurrent death | 0 | 1 | 0 | 0
Not completed — Other | 5 | 1 | 1 | 2
Not completed — Not treated | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set consisted of all enrolled subjects who received at least one dose of study drug, regardless of their eligibility to enter the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Adipocyte Tumors (ADI) | Leiomyosarcoma (LMS) | Synovial Sarcoma (SYN) | Other Types of Sarcoma (OTH) | Total
Number analyzed (Participants) | 37 | 40 | 19 | 31 | 127
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.1 (11.35) | 59.9 (12.69) | 43.7 (17.92) | 53.1 (15.21) | 54.4 (14.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 32 | 5 | 18 | 66
  Male | 26 | 8 | 14 | 13 | 61

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) at 12 Weeks
Description: PFS was determined from the Week 12 visit tumor scan and the participant's date of death. Progression was defined as complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), early death from any cause, or not assessable according to Response Evaluation Criteria In Solid Tumors (RECIST). CR defined as the loss of all target lesions. PR defined as ≥ 30% decrease in the sum of longest diameter (LD) of target lesions taking as reference the baseline sum LD. PD defined as ≥ 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since treatment started or the appearance of new lesions. SD defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum LD since treatment started. The number and percentage of successes were summarized by stratum and overall, together with 95% 2-sided confidence intervals (CIs) for the percentage of successes.
Time Frame: Week 12
Population: Efficacy evaluable set (EES) consisted of all registered, eligible subjects who had received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adipocyte Tumors (ADI) | Leiomyosarcoma (LMS) | Synovial Sarcoma (SYN) | Other Types of Sarcoma (OTH)
Number analyzed (Participants) | 32 | 38 | 19 | 26
Percentage of participants | 46.9 [29.1 to 65.3] | 31.6 [17.5 to 48.7] | 21.1 [6.1 to 45.6] | 19.2 [6.6 to 39.4]

2. Secondary Outcome: Overall Progression Free Survival
Description: Overall PFS was determined from any evidence that the participant had progressed, along with whether or not the participant was still alive at the end of the study. Tumors were evaluated every 6 weeks during treatment, and at least 4 weeks after the first observation of a complete or partial response. After discontinuation of study drug, participants without PD were re-evaluated every 12 weeks, unless a new anticancer therapy was started. Participants were considered as having progressed if they were classed as PD at Week 12, or had a best overall response (BOR) of PD, or had a date of progression, if they discontinued due to PD, died due to PD, or if the PI had recorded a date of progression. A participant was determined progression free if they were alive without PD at the time of study cut-off. The number and percentage of successes were summarized by stratum and overall, together with 95% 2-sided CIs for the percentage of successes.
Time Frame: First dose of study drug to the date of disease progression or date of death, whichever occurs first, or date of study cut-off 28 Jun 2012, up to 5.5 years
Population: EES
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Adipocyte Tumors (ADI) | Leiomyosarcoma (LMS) | Synovial Sarcoma (SYN) | Other Types of Sarcoma (OTH)
Number analyzed (Participants) | 32 | 38 | 19 | 26
Days | 82 [44 to 175] | 88 [69 to 114] | 81 [43 to 101] | 72 [42 to 87]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants in the analysis set who had a BOR of CR or PR based on RECIST v. 1.0 for target lesions. Tumors were assessed using x-rays, magnetic resonance imaging (MRI), or computed tomography (CT) scans, or both, as appropriate. ORR was documented and confirmed by two measurements taken at least 4 weeks apart. CR was defined as the disappearance of all target lesions. PR defined as ≥ 30% decrease in the sum of LD of target lesions taking as reference the baseline sum LD. Best overall response was derived using the same hierarchy as used when determining the PFS status at Week 12. No adjustments were made for participants who started further anticancer therapy prior to disease progression. 95% CIs were calculated using the exact method of binomial distribution. ORR = CR + PR
Time Frame: Date of first dose of study drug until documentation of CR or PR, or up to data cutoff 28 Jun 2012, up to approximately 5.5 years
Population: EES
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adipocyte Tumors (ADI) | Leiomyosarcoma (LMS) | Synovial Sarcoma (SYN) | Other Types of Sarcoma (OTH)
Number analyzed (Participants) | 32 | 38 | 19 | 26
Percentage of participants | 3.1 [0.1 to 16.2] | 5.3 [0.6 to 17.7] | 5.3 [0.1 to 26.0] | 3.8 [0.1 to 19.6]

4. Secondary Outcome: Clinical Response Benefit (CRB)
Description: CRB was defined as the percentage of participants with a BOR of CR or PR or SD as defined by RECIST, described previously. BOR was derived using the same hierarchy as used when determining the status at Week 12. No adjustments were made for participants who started further anticancer therapy prior to disease progression. 95% CIs were calculated using the exact method of binomial distribution. CRB = CR + PR + SD
Time Frame: Date of first dose of study drug to documentation of CR, PR, or SD, or until data cutoff date 28 Jun 2012, up to approximately 5.5 years
Population: EES
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adipocyte Tumors (ADI) | Leiomyosarcoma (LMS) | Synovial Sarcoma (SYN) | Other Types of Sarcoma (OTH)
Number analyzed (Participants) | 32 | 38 | 19 | 26
Percentage of participants | 59.4 [40.6 to 76.3] | 57.9 [40.8 to 73.7] | 47.4 [24.4 to 71.1] | 46.2 [26.6 to 66.6]

5. Secondary Outcome: Time to Onset of Response
Description: Time to onset of response could be calculated only if a participant achieved an objective response (BOR of CR or PR as defined previously). Participants who never achieved CR or PR were not included in the Kaplan-Meier survival estimates for the time to onset of response by strata. Given the small number of participants with these responses and the large variation in time to onset of response between participants, no comparison could be made among the strata.
Time Frame: Date of first dose of study drug to date of first documented CR or PR, or until data cutoff date 28 Jun 2012, up to approximately 5.5 years
Population: EES
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Adipocyte Tumors (ADI) | Leiomyosarcoma (LMS) | Synovial Sarcoma (SYN) | Other Types of Sarcoma (OTH)
Number analyzed (Participants) | 32 | 38 | 19 | 26
Days | 86 [NA to NA] — Not calculable (n=1) | 166 [120 to 211] | 77 [NA to NA] — Not calculable (n=1) | 42 [NA to NA] — Not calculable (n=1)

6. Secondary Outcome: Duration of Response
Description: Duration of response could be calculated only if a participant achieved a BOR of CR or PR, as defined previously. For consistency with the formula used by the European Organization for Research and Treatment of Cancer (EORTC), the duration was derived as "day of event minus day of first documented CR or PR" (one was not added to the calculation). Participants who were alive without documented progression had their duration of response censored at the day of last follow-up for progression. Participants who never achieved CR or PR were not included in the Kaplan-Meier survival estimates for the duration of response by strata. No adjustment was made for participants who started further anticancer therapy prior to disease progression.
Time Frame: Date of first documented CR or PR until the date of first document disease progression (or death), or up to data cutoff 28 Jun 2012, up to approximately 5.5 years
Population: EES
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Adipocyte Tumors (ADI) | Leiomyosarcoma (LMS) | Synovial Sarcoma (SYN) | Other Types of Sarcoma (OTH)
Number analyzed (Participants) | 32 | 38 | 19 | 26
Days | 418 [NA to NA] — Not calculable (n=1) | 129 [85 to 173] | 102 [NA to NA] — Not calculable (n=1) | 85 [NA to NA] — Not calculable (n=1)

7. Secondary Outcome: Overall Survival (OS)
Description: Participants still alive at the end of the study had their time to event censored at the day last known to be alive. Participants lost to follow-up were also censored at the date last known to be alive. 95% CIs for the percentage of participants still alive at the end of the study were presented as described for the primary endpoint, PFS at Week 12.
Time Frame: Date of first dose of study drug to date of death from any cause, or up to cut-off date of 28 Jun 2012, up to approximately 5.5 years
Population: EES
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Adipocyte Tumors (ADI) | Leiomyosarcoma (LMS) | Synovial Sarcoma (SYN) | Other Types of Sarcoma (OTH)
Number analyzed (Participants) | 32 | 38 | 19 | 26
Days | 363 [234 to 495] | 466 [392 to 697] | 293 [170 to 371] | 204 [149 to 312]

8. Secondary Outcome: Summary of Adverse Events (AEs)
Description: Treatment-emergent adverse events (TEAEs) and serious adverse events were reported. TEAEs are defined as an adverse event (AE) that emerged during treatment, having been absent at baseline or: reemerged during treatment, having been present at pretreatment (baseline) but stopped before treatment, or worsened in severity during treatment relative to the pretreatment state, when the AE was continuous. All AEs and SAEs were graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. A participant was counted only once within a System Organ Class (SOC) and preferred term (PT), even if the participant experienced more than one TEAE with a specific SOC and PT. Participants were summarized by treatment group according to the worst CTCAE grade assigned for each PT. Treatment-related TEAEs included TEAEs that were considered by the investigator to be possibly or probably related to study drug or TEAEs with a missing relationship.
Time Frame: Day 1 of study treatment until progressive disease, or up to cut-off date of 28 Jun 2012, up to approximately 5.5 years
Population: Safety analysis set included all participants who received at least one dose of study drug, regardless of their eligibility to enter the study.
Measure: Number; unit: Percentage of participants
Arm/Group | Adipocyte Tumors (ADI) | Leiomyosarcoma (LMS) | Synovial Sarcoma (SYN) | Other Types of Sarcoma (OTH)
Number analyzed (Participants) | 37 | 40 | 19 | 31
Percentage of participants
  TEAEs | 97.3 | 95.0 | 100.0 | 100.0
  Treatment-related TEAEs | 94.6 | 87.5 | 94.7 | 83.9
  TEAEs with CTCAE Grade 3 or 4 | 54.1 | 45.0 | 47.4 | 58.1
  Serious TEAEs | 37.8 | 30.0 | 36.8 | 45.2
  TEAEs leading to death | 2.7 | 5.0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious AEs were collected from time of signed consent until 30 days after last protocol treatment, up to approximately 5.5 years.
Description: Treatment-emergent adverse events (TEAEs) were reported and are defined as an AE that emerged during treatment, having been absent at baseline or: reemerged during treatment, having been present at pretreatment (baseline) but stopped before treatment, or worsened in severity during treatment relative to the pretreatment state, when the AE was continuous. All AEs and SAEs were graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Arm/Group | Adipocyte Tumors (ADI) | Leiomyosarcoma (LMS) | Synovial Sarcoma (SYN) | Other Types of Sarcoma (OTH)
Serious Adverse Events (participants affected / at risk) | 14/37 | 12/40 | 7/19 | 14/31
Other Adverse Events (participants affected / at risk) | 36/37 | 38/40 | 19/19 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adipocyte Tumors (ADI) (N=37) | Leiomyosarcoma (LMS) (N=40) | Synovial Sarcoma (SYN) (N=19) | Other Types of Sarcoma (OTH) (N=31)
General physical health deterioration (General disorders) | 2 | 2 | 1 | 0
Pyrexia (General disorders) | 2 | 1 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 2
Catheter site infection (Infections and infestations) | 1 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 3
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cerebral ischcaemia (Nervous system disorders) | 0 | 1 | 1 | 0
Anterior spinal artery syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Ureteric stenosis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Pelvic venous thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adipocyte Tumors (ADI) (N=37) | Leiomyosarcoma (LMS) (N=40) | Synovial Sarcoma (SYN) (N=19) | Other Types of Sarcoma (OTH) (N=31)
Fatigue (General disorders) | 26 | 30 | 13 | 20
Pyrexia (General disorders) | 8 | 9 | 6 | 4
Oedema peripheral (General disorders) | 6 | 9 | 2 | 5
Chest pain (General disorders) | 3 | 5 | 1 | 1
Chills (General disorders) | 4 | 0 | 2 | 0
General physical health deterioration (General disorders) | 2 | 21 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 2 | 1 | 1
Influenza like illness (General disorders) | 1 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 16 | 12 | 9 | 8
Constipation (Gastrointestinal disorders) | 6 | 14 | 6 | 8
Diarrhoea (Gastrointestinal disorders) | 9 | 12 | 4 | 5
Abdominal pain (Gastrointestinal disorders) | 11 | 7 | 4 | 7
Vomiting (Gastrointestinal disorders) | 11 | 7 | 3 | 5
Stomatitis (Gastrointestinal disorders) | 5 | 9 | 3 | 7
Dyspepsia (Gastrointestinal disorders) | 2 | 8 | 0 | 3
Abdominal distension (Gastrointestinal disorders) | 4 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 3
Flatulence (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Oral pain (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 17 | 16 | 7 | 6
Dizziness (Nervous system disorders) | 6 | 12 | 1 | 8
Headache (Nervous system disorders) | 7 | 8 | 1 | 7
Dysgeusia (Nervous system disorders) | 6 | 7 | 3 | 3
Peripheral motor neuropathy (Nervous system disorders) | 3 | 3 | 2 | 3
Neuralgia (Nervous system disorders) | 1 | 2 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 11 | 10 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 9 | 6 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 16 | 24 | 10 | 11
Exfoliative rash (Skin and subcutaneous tissue disorders) | 2 | 6 | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 5 | 2 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 7 | 6 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 5 | 4 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 5 | 5 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 11 | 11 | 16
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 3
Weight decreased (Investigations) | 11 | 12 | 7 | 4
Weight increased (Investigations) | 5 | 4 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 9 | 15 | 6 | 9
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 1 | 5 | 3 | 3
Cystitis (Infections and infestations) | 0 | 3 | 0 | 3
Pharyngitis (Infections and infestations) | 2 | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 2 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 2
Herpes zoster (Infections and infestations) | 0 | 1 | 1 | 0
Oral infection (Infections and infestations) | 0 | 0 | 1 | 0
Skin candida (Infections and infestations) | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 6 | 5 | 0 | 4
Anxiety (Psychiatric disorders) | 2 | 3 | 3 | 4
Depression (Psychiatric disorders) | 3 | 3 | 1 | 4
Confusional state (Psychiatric disorders) | 1 | 2 | 0 | 1
Hypertension (Vascular disorders) | 3 | 2 | 1 | 1
Hypotension (Vascular disorders) | 0 | 1 | 2 | 2
Embolism (Vascular disorders) | 1 | 1 | 1 | 0
Flushing (Vascular disorders) | 0 | 3 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 0
Vena cava embolism (Vascular disorders) | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 1 | 3 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 4 | 1 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 3 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 2
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Ocular surface disease (Eye disorders) | 3 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 2 | 0 | 0
External ear pain (Ear and labyrinth disorders) | 2 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other